CLINICAL TRIAL: NCT00788502
Title: Stress Reduction During In Vitro Fertilization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SU-11052008-1334; 15402 (Other: Stanford University IRB)
Record Dates: First submitted 2008-11-06; First posted 2008-11-11 (Estimated); Last update posted 2022-06-09 (Actual); Status verified 2022-06

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility | interventions — Touch; Desensitization, Psychologic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Healing Touch (Experimental): Healing Touch (HT) is a gentle form of energy balancing work that promotes relaxation. Subjects in this arm will receive three one-hour sessions of Healing Touch during the first two weeks of their IVF cycle.
  Interventions: Behavioral: Healing Touch
- Desensitization Therapy (Experimental): Desensitization Therapy is a quasi-desensitization procedure where subjects meet with a therapist and generate a list of stressful thoughts and a list of neutral thoughts. Subjects in this arm will receive three one-hour sessions of Desensitization Therapy during the first two weeks of their IVF cycle.
  Interventions: Behavioral: Desensitization Therapy
- Standard Care (No Intervention): Subjects in this arm will receive no therapeutic intervention.

INTERVENTIONS:
Behavioral: Healing Touch
  Arms: Healing Touch
Behavioral: Desensitization Therapy
  Arms: Desensitization Therapy

SUMMARY:
The goal of this study is to determine the effect of Healing Touch (HT) on the stress, anxiety, and self-efficacy experiences of women undergoing in vitro fertilization (IVF) in a randomized, controlled design. HT is a gentle, non-invasive form of energy-balancing work that promotes relaxation.

DETAILED DESCRIPTION:
Once enrolled, each participant will be randomized to one of three groups: the Healing Touch (HT) treatment arm, the Desensitization Therapy (DT) arm, or the no-intervention arm.

Subjects in Group 1 will receive three, 45-minute HT sessions during the first two weeks of their IVF cycle prior to oocyte retrieval. Group 2 will receive three, 45-minute DT sessions during the first two weeks of their IVF cycle prior to oocyte retrieval. Group 3 will receive no intervention. Subjects in Group 3 will be offered two HT sessions after completing study participation.

All subjects and their partners will be asked to complete the Spielberger State Trait Anxiety Inventory (STAI), the Perceived Stress Scale (PSS) and the Infertility Self-Efficacy Scale (ISES) at three time points: 1) baseline 2) one day prior to oocyte retrieval and 3) 5-7 days post embryo transfer. In addition, subjects in all groups will complete a short pre-study questionnaire to assess expectation of therapeutic effect, and subjects in the two intervention groups will complete a short post-study questionnaire to evaluate their treatment experience. Demographic and pregnancy outcome data will be collected for all subjects.

ELIGIBILITY:
Inclusion Criteria:-Age <43

* FSH <= 14
* About to enter an IVF cycle at the Stanford Fertility and Reproductive Medicine Center
* Planning a transfer of their own fresh embryos during this cycle
* Speak and read English fluently
* Not planning to use concomitant energy work interventions (HT, Reiki, QiGong, acupuncture)during the IVF cycle.

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2008-10; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Spielberger State Trait Anxiety Inventory | 30 days

SECONDARY OUTCOMES:
Perceived Stress Scale | 30 days
Infertility Self-Efficacy Scale | 30 days
Pregnancy outcome | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Kathy Turner RN, NP, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States